CLINICAL TRIAL: NCT07053241
Title: The Effect of the Web-Based Gamified Application Developed for Post-Total Knee Replacement Surgery Care on Functional Results and Recovery Conditions
Brief Title: The Effect of the Web-Based Gamified Application on Functional Results and Recovery Conditions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Cafer Özdemir, Principal Investigator, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: AAU-4293-2020
Record Dates: First submitted 2025-01-06; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Recovery; Functional Outcome
Keywords: Postoperative recovery; Functional outcome; Total knee arthroplasty; Surgical nursing; Education programme; Rehabilitation; Gamification; Mobile application; Web-based; Randomized controlled trial
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Single-blind pre-test-post-test measurement, follow-up, and single-center randomized controlled design.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The intervention and control groups will be given an explanation of the study independently after discharge. Both groups will have access to the application. However, only the intervention group will have access to the game module.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Game Module + Education Booklet Module
  Interventions: Device: Game-App-KNEE
- Control Group (Placebo Comparator): Education Booklet Module
  Interventions: Other: Control group (standart care)

INTERVENTIONS:
Device: Game-App-KNEE — * In the outpatient clinic phase of the study, the purpose of the study will be explained to individuals who meet the inclusion criteria.
  * The mobile-compatible web-based gamified application created for individuals included in the intervention group will be downloaded to patients' phones in the outpatient clinic phase and information will be provided on how to use the application, and the training will be repeated if they have questions.
  * Individuals in the intervention group will be able to access both the education module in PDF format and the game module containing the gamified education program for three months in the application.
  * In-app reminder messages will be sent to individuals to actively use the application. (We missed you today, warrior, where are you, let's finish this job, etc.)
  * Whether the application is actively logged in, how long it is in the application, and the level of success in the game will be monitored by the researcher from the administrator panel.
  Arms: Intervention Group
Other: Control group (standart care) — Description: In the outpatient clinic phase of the study, the purpose of the study will be explained to individuals who meet the inclusion criteria. -An application will be installed on the phones of individuals included in the control group during the outpatient clinic phase. -In the first information phase, individuals will be registered to the system with their username and password by the researcher via their smartphones or tablets and will be allowed to enter the application. Considering that the participant may forget their username and password, a 'forgot my password' button will be added. -Individuals in the control group will only be able to access the training module in PDF format for three months.
  Arms: Control Group

SUMMARY:
The aim of this clinical trial is to determine the effect of a mobile-compatible web-based gamified application (Game-App-KNEE) developed for post-operative care of total knee replacement (TKA) surgery on functional outcomes and recovery status.

Based on this, the hypotheses of our project are; In the intervention group where the mobile-compatible web-based gamified application to be developed for the home care of individuals undergoing TKA due to osteoarthritis is applied, compared to the control group; Hypothesis 1 (H1): After the application of Game-App-KNEE, the functional levels of individuals in the intervention group are higher than the control group.

Hypothesis 2 (H1): After the application of Game-App-KNEE, the post-operative recovery levels of individuals in the intervention group are higher than the control group.

Participants:

Receive the game module application (intervention group) or only the educational booklet (control group) every day for 3 months after discharge Visit the clinic every 1st and 3rd month for check-ups and tests.

DETAILED DESCRIPTION:
METHOD This project is planned in two phases. In the first phase, the development of the Game-App-KNEE is intended to enable individuals undergoing Total Knee Prostheses (TDP) to manage their postoperative process. Additionally, it aims to evaluate the content of the educational program to be integrated into the application, as well as the design of the sections that will be included in the application, and to assess the technical suitability and usability of the application.

In the second phase, a randomized controlled study is planned to determine the effect of the mobile-compatible web-based gamified application, which integrates the educational program, on individuals' functional outcomes and recovery status.

FIRST PHASE Creation of the Mobile-Compatible Web-Based Gamified Application The design process of the mobile-compatible web-based gamified application consists of specific stages. These stages are presented in Table 1.

Table 1. Design Process of a Mobile-Compatible Web-Based Gamified Application Creation of the Educational Program Content to be Included in a Mobile-Compatible Web-Based Gamified Application

* Literature Review
* Preparation of Educational Content to be Implemented
* Obtaining Expert Opinions Using the Lawshe Technique
* Evaluation of Educational Content Using the Readability Formula
* Updating Educational Content Based on Expert and Patient Opinions and the Readability Formula
* Finalizing the Content Template Design of a Mobile-Compatible Web-Based Gamified Application
* Conducting Player Analyses for 6 Patients from the Target Patient Group Planned for the Application
* Preparing the Gamification Template Based on the Results of the Player Analyses Development of a Mobile-Compatible Web-Based Gamified Application and Conducting a Pilot Study
* Design of the Application Logo
* Design of the Application Interfaces
* Integration of the Gamification Template into the Program
* Transfer of Interfaces to the Mobile Application and Testing of the Application
* Evaluation of the System Using the System Usability Scale (SUS) in Three Patients Who Underwent Total Knee Prosthesis Surgery

Preparation of a Mobile-Compatible Web-Based Gamified Application for Use -Updating the Application Based on Feedback from Patients and Issues Experienced

IP 1. Development of the Educational Program to be included in the Mobile-Compatible Web-Based Gamified Application In the preparation phase of the educational program for the mobile-compatible web-based gamified application, the educational content will first be created, and then this prepared educational content will be evaluated.

IP 1.1 Creation of the Educational Program Content to be included in the Mobile-Compatible Web-Based Gamified Application During the creation of the educational content, various databases such as PubMed, Web of Science, Cochrane Library, Science Direct, and EBSCO, as well as the websites and guidelines of national/international scientific associations, will be scanned to identify studies related to the home care process and self-care following Total Joint Replacement (TJR), along with the educational needs. The literature review, along with insights from experts and patients, will guide the researcher in developing the educational content to be integrated into the mobile-compatible web-based gamified application. A comprehensive literature review has been conducted using the identified keywords for the subject headings of the educational program content to be included in the mobile-compatible web-based gamified application. The keywords used in the literature review include "postoperative recovery, functional outcomes, total knee prosthesis, surgical nursing, educational program, rehabilitation, gamification, mobile application, web-based, randomized controlled trial." The headings related to the content of the educational program are presented in Table 2.

Table 2. Content of the Training Program GENERAL INFORMATION What is osteoarthritis? What is total knee replacement surgery? What are the possible complications and adverse conditions that may develop after total knee replacement? When should you seek emergency medical attention? HOME REHABILITATION PROCESS What should you pay attention to in pain management at home? What should you consider in physical therapy and home exercises? What should you be mindful of in addressing self-care needs and daily activities? What should you focus on in surgical wound management? What should you ensure when maintaining a proper nutrition regimen? What should you consider in establishing a sleep routine? What should you pay attention to in preventing complications and adverse situations? Prevention of thrombosis (Embolism) Prevention of infection Prevention of falls Exercises IP 1.2 Evaluation of the Content of the Training Program The first draft of the training program content to be integrated into the mobile-compatible web-based gamified application to be developed was presented to the Thesis Monitoring Committee members and the suggested corrections were made. The training content, which was ready for expert opinion, was submitted to expert opinion via e-mail. Experts evaluated each topic and content with the expert opinion form prepared by the researcher. Opinions and suggestions about the relevant sections of the training program were obtained from the experts through this form. The experts did not recommend the removal of any section. The evaluation of expert opinions was analyzed with the Kendall Concordance Coefficient. Opinions were received from a total of ten experts (Appendix-1), from the fields of Surgical Diseases Nursing (n=6), Internal Medicine Nursing (n=1), Orthopedics and Traumatology Department (n=2), Physiotherapy and Rehabilitation Department (n=1). According to the analysis, it was determined that the agreement between the experts was significant (W= 0.364, p<0.05). The use of the program was found appropriate after expert opinions and the Kendall coefficient. Later, the difficulty level of the application content was determined by the researcher using the "Ateşman Readability Formula" (Ateşman, 1997). The readability score of the training content was calculated as 66.6 (Medium Difficulty).

• Atesman Readability Formula The tool is used to evaluate the readability of text content for each patient. Ateşman's Readability Formula was developed by Ateşman in 1997. Ateşman, who claims that the formula developed by Flesch (Farr et al., 1951) is the most suitable formula for the unique structure of Turkish, states that this formula was created for English texts and that the formula shaped on the variables of sentence length and word length should be adapted. Ateşman adapted Flesch's formula to Turkish as a result of various applications and calculations he made.

The formula is as follows:

Readability number = 198.825 - 40.175. X1 - 2.610. X2 X1= Average word length in syllables X2= Average sentence length in words (Ateşman, 1997). In this formula, the first 100 words in the text examined are evaluated to find the readability number. The total syllable length of these 100 words taken into consideration is divided by 100 to find X1, and the 100 words are divided by the number of sentences to find X2. These values are written in their places in the formula to obtain the readability score of the text. The scores obtained as a result of this formula are classified as; 90-100 as "Very Easy", 70-89 as "Easy", 50-69 as "Medium Difficulty", 30-49 as "Difficult" and 1-29 as "Very Difficult" readability level (Çoban, 2014).

IP 2. Creation of Mobile Compatible Web-Based Gamified Application Template When creating the template of the mobile-compatible web-based gamified application, first of all, player analyses of the group to be included in the sample were conducted and the gamification template was created with the data obtained from these analyses.

IP 2.1. Performing Player Analyses for Mobile Compatible Web-Based Gamified Application Patients will have both an entertaining experience and access the information they want with the information provided in the mobile-compatible web-based gamified application. In the schematization of the mobile-compatible web-based gamified application, dynamics, elements, and components were taken into consideration and a survey was applied to 6 individuals who had total knee prostheses to determine the player types of the target audience who will use the program (Akgün & Topal, 2018). As a result of the obtained data, player types were analyzed (persona analysis) by the researcher.

IP 2.2. Preparation of Mobile Compatible Web-Based Gamified Application Template A mobile-compatible web-based gamified application template was prepared in line with the player analyses.

IP 3. Development of Mobile Compatible Web-Based Gamified Application Game-App-KNEE will be developed according to the gamification template prepared in line with the dynamics, mechanics, elements, and gamification framework in the gamification pyramid.

IP 3.1 Logo, Interface, Graphic Design, and Integration of Mobile-Compatible Web-Based Gamified Application The content of the training program includes pain management, physical therapy, and home exercises, as well as prevention of complications, self-care, wound management, sleep management, and nutrition management. After the content of the training program is created and the financial processes are completed, the logo, user interfaces, and graphic design of the application will be designed by an authorized software company and an expert team. The colors of the application and where the content will be will be decided in this section. Question templates were created by the researcher in line with the information specific to each area in the training program (Appendix 3). In addition to the question templates, the application content will be supported by videos, animations, photographs, and pictures created by the researcher or with the help of artificial intelligence. The cost and legal status of the mobile-compatible web-based gamified application software will also be evaluated in the first stage.

The cost of a mobile-compatible web-based gamified application varies depending on the type of content (video, animation, photo, image). Various gamification elements will be added to the application content and the cost will increase as elements are added.

IP 4. Implementation of the Pilot Study of the Research The mobile-compatible web-based gamified application, whose software process has been completed, will be tested by experts, researchers, and patients who have undergone knee replacement surgery in order to evaluate its operation and detect and correct errors. In order to evaluate the usability of the system, the System Usability Scale (SUS), developed by Brooke in 1996 (Brooke, 1996) and adapted to the Turkish society by Demirkol and Seneler, and whose validity and reliability have been performed, will be used (Demi̇rkol & Seneler, 2018). As a result of the feedback received, problems in the application will be determined and technical support will be received.

A pilot study is planned to be conducted with three patients who have undergone total knee replacement surgery before the research to test the application and evaluate its comprehensibility. The patients included in the pilot study will not be included in the study. After the pilot study, feedback will be received from the patients regarding the suitability, content, structure, language, images, font size, and visual and audio quality of the application and the detected problems will be corrected. At this stage, the processes regarding all corrected, changed, added, or removed information will be completed and the application will be finalized. The aim will be to update and improve the application.

SECOND STAGE IP 5. Conducting a Randomized Controlled Trial The randomization processes of this study were prepared in accordance with the guide created by CONSORT for Randomized Controlled Trials (Cuschieri, 2019).

Type of Study: In this phase of our project, a single-blind, pre-test post-test measurement, observational, and single-center randomized controlled study is planned. An application will be made for Clinical Trials registration.

Place and Time of Study: The study will be conducted at the Antalya City Hospital Orthopedics and Traumatology Clinic. When routine practices specific to orthopedic surgery at the Health Sciences University Antalya City Hospital are examined, the patient's suitability for surgery is first evaluated. In this direction, the patient is evaluated by the orthopedist and anesthesiologist and the necessary tests are performed. After the evaluation, the patient is given a date for surgery. The patient comes one day before the surgery or in the morning of the surgery day and gets admitted, depending on the availability of the clinic and himself. Patients usually stay in the clinic for an average of three days after surgery. Patients come for a check-up within 10 days to a month after discharge. Afterward, physical therapy is recommended to the patient. The patient is not followed up after discharge. Only verbal information is given to the patients by the doctor and nurse during discharge. It is planned to complete the research data in 24 months between 10.08.2024 and 10.08.2026 after obtaining permissions.

Universe and Sample of the Research: The universe of the research will consist of patients between the ages of 18-65 who underwent elective TDP surgery with spinal anesthesia technique due to osteoarthritis diagnosis at Antalya Education and Research Hospital and Antalya City Hospital Orthopedics Clinic and who did not develop any complications until discharge. The sample of the research will consist of patients who meet the inclusion criteria of the research.

Sample Size The G Power 3.1 analysis program was used to calculate the sample size of the study. Power is the probability of capturing the difference between the two groups of the study. The power is desired to be at least 80%. Type 1 error is defined as finding a difference in the study result when there is no real difference between two applications based on H0, and the p-value indicates the probability of type 1 error. In order for a statistically significant difference to exist, the p-value must be below 0.05 (Campbell et al., 2010). According to the power analysis conducted in line with a technology-based study on TDP patients in the literature (P. Huang et al., 2017) for the sample size in this study; it was determined that the minimum sample size of 21 interventions and 21 control groups was sufficient for large effect size (d = 0.78) for 80% power and 0.05 error.

In order to strengthen the research results, increase its reliability, and prevent losses during the research, it is planned to be conducted with 54 patients, 27 in the intervention group and 27 in the control group, as a result of a 30% increase.

Randomization The study plans to control selection bias by performing random assignment and concealing randomization. Randomization involves randomly assigning participants included in the study to the intervention and control groups. In this way, each subject enters any group with equal and known probability (Tabachnick & Fidell, 2013). In the study, randomization will be performed in order to provide equal samples for the intervention and control groups using a pre-test and post-test control group design. In order to provide equal samples for both groups in the randomization to be performed, the "stratified randomization method" will be used. Patients will be randomized stratified according to age and body mass index. It is stated that age is a determinant of complications and functional outcomes (Passias et al., 2020) and that body mass index increases the risk of revision and slows down recovery (Tohidi et al., 2018). In the stratified randomization stage, numbers will be generated in a computer environment via https://www.randomizer.org/ and the generated numbers will be placed in opaque, closed envelopes. The randomization stage will be performed by a person independent of the research team. The researcher will determine whether the patient is in the intervention or control group by opening the envelope given by the person performing the randomization. After randomization, the homogeneity between the intervention and control groups will be determined by number, percentage, chi-square, and t-test. In order to ensure homogeneity, when three patients are reached in the intervention and control groups, the groups will be examined by number, percentage, chi-square, and t-test based on the pre-tests of the individuals.

Blinding and Preventing Bias Randomization will be performed in the study to prevent selection bias. It is planned to blind the patients and the statistician. Blinding the researcher will not be possible. Since the patients do not know which group they will be assigned to, patient blinding is considered possible. Separate informed consent forms will be prepared for individuals in the control group and those in the intervention group, and in order to ensure blinding, individuals in the control group will also be given a password to enter the application, but individuals in the control group will only be able to access the training module in the application. Data related to the scales (post-test) will be coded as 'A' and 'B' without specifying the intervention and control groups. The analysis of the coded data in terms of groups will be carried out by the statistician. After the statistical analyses are performed, the coding for the intervention and control groups will be explained. It is planned to control statistical bias with this blinding technique.

IP 5.1 Collection of Research Data The Introductory Information Form, System Usability Scale (SUS), WOMAC Osteoarthritis Index (Western Ontario and McMaster Universities Osteoarthritis Index), and Postoperative Recovery Index (PoRI) will be used in the data collection process of the research. All patients who meet the inclusion criteria will be included in the research until the sample size is reached, and the patients included in the research will be informed about the research process and their written and verbal consent will be obtained.

Intervention Group In the outpatient clinic phase of the study, the purpose of the study will be explained to individuals who meet the inclusion criteria.

The mobile-compatible web-based gamified application created for individuals included in the intervention group will be downloaded to patients' phones in the outpatient clinic phase and information will be provided on how to use the application, and the training will be repeated if they have questions.

In the first information phase, individuals will be registered to the system by the researcher with their username and password via their smartphones or tablets and will be allowed to enter the application. Considering that the participant may forget their username and password, a 'forgot my password' button will be added.

Individuals in the intervention group will be able to access both the education module in PDF format and the game module containing the gamified education program for three months in the application.

In-app reminder messages will be sent to individuals to actively use the application. (We missed you today, warrior, where are you, let's finish this job, etc.) Whether or not the application is actively logged in, how much time is left in the application, and the level of success in the game will be monitored by the researcher from the admin panel.

The use of the mobile-compatible web-based gamified application will be reinforced with individuals in the intervention group who come to the outpatient clinic on the 15th day after the surgery, and detailed information will be repeated to the individuals about the parts they have difficulty using the application.

Control Group In the outpatient clinic phase of the study, the purpose of the study will be explained to individuals who meet the inclusion criteria.

The application will be downloaded to the phones of the individuals included in the control group during the outpatient clinic phase.

In the first information phase, the individuals will be registered to the system with their username and password by the researcher via their smartphones or tablets and they will be allowed to enter the application. Considering that the participant may forget their username and password, a 'forgot my password' button will be added.

Individuals in the control group will only be able to access the training module in PDF format for three months.

Ethics Committee Approval Permission for the research was obtained from the Akdeniz University Faculty of Medicine Clinical Research Ethics Committee (Decision No: KAEK-572, Date: 19.07.2023). Necessary permissions were obtained from Antalya City Hospital (Document No: E-98360293-604.01-249242699) and Antalya Provincial Health Directorate (Document No: E-98360293-604.01-249375909) where the research will be conducted. After the purpose of the study is explained to the individuals who will be included in the research sample, written and verbal consent will be obtained from the individuals who voluntarily accept the research. The research data will be collected in accordance with the Declaration of Helsinki after the purpose of the research is explained to the individuals.

*Study Variables Dependent Variables: Functional Outcomes, Postoperative Recovery Status Independent Variables: Mobile Compatible Web-Based Gamified Application IP 5.2 Completion of Statistical Analyses of the Study, Evaluation of Research Results The Statistical Package for Social Science (SPSS) 26.0 (IBM Corporation, Armonk, NY, USA) package program will be used in the analysis of the data obtained as a result of the study. The sample size and power analysis of the data were determined using the G*Power (v. 3.1) program. In this study conducted to determine the effect of individuals who underwent total knee arthroplasty on functional outcomes and postoperative recovery status after the application, the structure of the score distributions of the intervention and control groups in the relevant independent variable will be examined first. Before the analyses, the conformity of the continuous variables to the normal distribution in the groups will be checked with the Kolmogorov Smirnov (KS) and Shapiro-Wilks (S-W) tests. If the p-values of the obtained test results are greater than 0.05, the distribution in question will be accepted as normal. Another method used to decide on the distribution structure is the kurtosis and skewness coefficients of the distribution. If these coefficients are between -1 and 1, the distribution will be assumed to be normal (Büyüköztürk et al., 2000a). Finally, the kurtosis and skewness Z values were used to decide on the structure of a score distribution. If these values are between -1.96 and 1.96, the distribution will be considered normal (Çelik, 2023; George & Mallery, 2010). Distributions that meet at least two criteria from the above-mentioned methods will be accepted as normal distributions. In cases where the data are suitable for a normal distribution, parametric tests will be used, and in cases where it is not, nonparametric tests will be used to analyze the descriptive statistics of the variables. The descriptive statistics of the variables will be presented with a number (n), percentage (%), mean (x̄), standard deviation (ss), median, interquartile range (IQR), and minimum-maximum values. Whether there is a difference in descriptive data between the intervention and control groups will be determined using chi-square analysis for categorical variables. If all subgroups of independent variables with two subgroups show normal distribution, an independent groups t-test will be used, and if at least one subgroup does not show normal distribution, Mann Whitney U test will be used. If all subgroups of independent variables with more than two subgroups show normal distribution, one-way analysis of variance (ANOVA) will be used, and if at least one subgroup does not show normal distribution, the Kruskal Wallis H test will be used. If the comparison of time-dependent (pretest-follow-up-posttest) score changes within the groups shows normal distribution, a dependent groups t-test will be applied, and if it does not show normal distribution, a signed ranks test will be applied. Intention to Treat (ITT) analysis will be performed for missing data in the evaluation of the research results. In completing the missing data in the post-tests, the worst-case scenario will be considered and missing data will be completed (Çelik, 2023; Günüşen & Üstün, 2009). In the next stage of the study, mixed measures analysis of variance will be applied to test the effectiveness of the intervention, in which group-time main effects and joint effects are tested. The eta squared (η2) value will be calculated to evaluate the effect size. The effect size (η2) is defined as weak if it is less than 0.1, moderate if it is 0.6, and large if it is greater than 0.14 (Büyüköztürk et al., 2000b). The correlation between the scales was tested with Pearson correlation analysis. The obtained data were evaluated at a significance level of p<0.05 at a confidence interval of 95%. Finally, simple and multiple linear regression analysis will be applied to determine whether the functional results and postoperative recovery status mean scores are predictive of each other (Çelik, 2023).

ELIGIBILITY:
Inclusion Criteria:

* Must be able to read and write Turkish
* Must have internet access
* Must have a mobile compatible smartphone (IOS, Android)
* Must be able to use a smartphone
* Must be between the ages of 18-65

Exclusion Criteria:

* Having vision or hearing problems
* Having a mental illness
* Performing bilateral surgery
* Applying general anesthesia
* Having emergency surgery
* Revision surgery during the follow-up period
* Wanting to leave the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Functional Results | preoperative period, 1st month postoperatively, 3rd month postoperatively
  WOMAC is a valid and reliable index widely used for the evaluation of patients with osteoarthritis. It is a recommended measure for osteoarthritis studies by the Rheumatology Clinical Trials Outcome Measures (OMERACT). The WOMAC Osteoarthritis Index, the validity and reliability of which was performed in Turkey, consists of three sub-dimensions and 24 questions questioning pain, stiffness and physical function. The maximum scores that can be obtained from the index are 20 for the pain sub-group, 8 for stiffness and 68 for physical function. The total Cronbach alpha coefficients for the three sub-dimensions at Time 1 and 2 were determined as pain: 0.75, 0.81; stiffness: 0.71, 0.76; physical function: 0.94, 0.96. High scores indicate increased pain and stiffness and deterioration in physical function.
Postoperative Recovery Status | the day after surgery, 1st month postoperatively, 3rd month postoperatively
  The Postoperative Recovery Index, tested for validity and reliability, consists of 37 items. It has 5 sub-dimensions: psychological symptoms, physical activities, general symptoms, bowel and appetite symptoms. The scores of the items in the sub-dimensions are added up, their means are calculated, and the sub-dimension scores are determined. For the total PoRI score, all 37 items are added up and their means are calculated. High scores from the index indicate that there are more problems in post-operative recovery, while low scores indicate that post-operative recovery is easier. The internal consistency Cronbach's alpha coefficient of the original scale was determined as 0.95. The internal consistency Cronbach's alpha coefficient of the scale, whose Turkish validity and reliability were performed , was determined as 0.97. In addition, it was determined that the five-factor structure of PoRI-TR, which

CONTACTS AND LOCATIONS:
Overall Officials: Ebru KARAZEYBEK, Study Director — Akdeniz University; Sadullah TURHAN, Study Director — Mİnİstry of Health of the Republıc of Türkiye
Locations (1):
- Akdeniz University, Antalya, Konyaaltı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Sharing is planned because the study is a doctoral thesis.